CLINICAL TRIAL: NCT06563882
Title: Postural Management of Hyperkyphosis to Improve Motor Performance and Pulmonary Function in Cardiac Rehabilitation Patients
Brief Title: Postural Management of Hyperkyphosis in Cardiac Rehab Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Collaborators: Zinman College of Physical Education and Sports Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0172-23HMO
Record Dates: First submitted 2024-05-04; First posted 2024-08-21 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Hyperkyphosis
Keywords: Home-based program; Graded exercise test; Spirometry; Flexicurve ruler; Six-minute walk test; Posture; Kyphosis index; Physical functional capacity; TUG test
MeSH Terms: conditions — Kyphosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Home-based exercise program (Experimental): Intervention Group: Hyperkyphotic participants will participate in a home exercise program designed to improve thoracic spine and shoulder mobility and flexibility, while also strengthening spine extensor muscles, alongside a cardiac rehabilitation exercise program. The home-based program will include six exercises to be performed three times a week over a period of 12 weeks.
  Interventions: Other: Home-based exercise program
- Cardiac rehabilitation exercise program - Hyperkyphosis (Other): Control Group: Hyperkyphotic participants will participate in a 12-week cardiac rehabilitation exercise program, consisting of two one-hour sessions per week at the cardiac rehabilitation center. These sessions will include aerobic activity along with a variety of resistance, flexibility, and balance exercises.
  Interventions: Other: No intervention
- cardiac rehabilitation exercise program - without hyperkyphosis (Other): Control Group: Participants without hyperkyphosis will participate in a 12-week cardiac rehabilitation exercise program, consisting of two one-hour sessions per week at the cardiac rehabilitation center. These sessions will include aerobic activity along with a variety of resistance, flexibility, and balance exercises.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: Home-based exercise program — The program will comprise of six exercises aimed at improving the mobility of the thoracic spine and shoulders, strengthening the extensor muscles of the spine, and enhancing the flexibility of the chest and anterior shoulders. Progression within the program will involve increasing exercise duration or repetitions/sets, along with implementing postural corrections in compound exercises. Participants will be instructed to perform the exercises at least three times a week.
  To heighten participants awareness of their daily posture, they will receive a daily scheduled message via WhatsApp reminding them to focus on their posture. Once a week, participants will be asked to submit a home exercise tracking report to monitor their adherence to the program. Additionally, exercises execution will be reviewed every two weeks, and adjustments to the program will be made accordingly.
  Arms: Home-based exercise program
Other: No intervention — No intervention
  Arms: Cardiac rehabilitation exercise program - Hyperkyphosis; cardiac rehabilitation exercise program - without hyperkyphosis

SUMMARY:
The goal of this clinical trial is to evaluate the efficacy of a home-based exercise program in managing hyperkyphosis, and its impact on physical performance and pulmonary function among cardiac rehabilitation patients.

The primary research question is: Can a home-based kyphosis-specific exercise program reduce thoracic hyperkyphosis and improve physical ability in cardiac patients undergoing cardiac rehabilitation? The study will consist of three groups: 1) Hyperkyphotic participants undergoing a 12-week exercise program at home, alongside a cardiac rehabilitation exercise program, 2) Hyperkyphotic participants solely undergoing cardiac rehabilitation exercise program, and 3) Participants without hyperkyphosis solely undergoing cardiac rehabilitation exercise program.

The groups will be evaluated based on measurements of kyphosis index, physical performance and spirometry at the beginning, after 6 weeks, and upon completion of the 12-week program.

ELIGIBILITY:
Inclusion Criteria:

* Heart patients who will be admitted for cardiac rehabilitation at Hadassah - Mount Scopus Hospital
* Normal stress test results.
* Independent mobility.
* Stable hemodynamic and respiratory status.
* Ability to speak and read basic Hebrewץ
* Ability to watch videos on a mobile phone or computer.
* Not receiving any other forms of physical therapy or physical treatment.

Exclusion Criteria:

* Presence of unstable angina.
* Neurological disorders or mental illnesses that interfere with communication.
* Movement disorders due to neurological disease.
* Severe orthopedic limitations hindering the execution of motor exercises.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2024-04-21 (Actual); Primary Completion 2025-05-02 (Actual); Study Completion 2025-05-02 (Actual)

PRIMARY OUTCOMES:
Degree of Kyphosis | Assessment will occur at baseline, after 6 weeks, and upon completion of the 12-week program.
  This measure will be obtained using a 60-centimeter flexicurve ruler, placed over the subject's back, from the C7 spinous process down to the T12 spinous process. Once attached to the back, the flexicurve molds according to its shape, allowing tracing of the thoracic curve onto paper. Maximum width and length measurements are then taken of the curve in centimeters in order to calculate the kyphosis index. Kyphosis index is calculated as the ratio of thoracic width to thoracic length. A higher index value indicates a greater degree of kyphosis, with values exceeding 13 considered hyperkyphosis. Assessment will occur at the program's start, after 6 weeks, and upon completion of the 12-week program.

SECONDARY OUTCOMES:
Maximum Metabolic Equivalents (METs) | The measurement will be taken at baseline and upon completion of the 12-week program.
  This measure represents the total workload achieved during a symptom-limited graded exercise test in order to assess the subject's cardiovascular exercise capacity. The METs score will be calculated using a validated computerized algorithm. The test will be performed on a treadmill, with the workload progressively increasing every 2-3 minutes (depending on the chosen protocol). The test protocol will be determined based on the participant's age, overall physical fitness level, and any orthopedic limitations. During the test, the electrical activity of the heart will be monitored using an electrocardiogram (ECG) for diagnostic purposes, such as the detection of myocardial ischemia (e.g., ST-segment depression). The test will be terminated when the participant reaches or exceeds 85% of the maximum predicted heart rate, when the participant indicates an inability to continue, or if there are any clinical symptoms, abnormal findings in the ECG, or abnormal physiological responses.
Peak Heart Rate | The measurement will be taken at baseline and upon completion of the 12-week program.
  The maximum heart rate attained during a graded exercise test.
Peak Systolic and Diastolic Blood Pressure | The measurement will be taken at baseline and upon completion of the 12-week program.
  The maximum systolic and diastolic blood pressure measured during a graded exercise test.
Distance covered in a six-minute walk test | The test will be conducted at baseline, after 6 weeks, and upon completion of the 12-week program.
  The Six-Minute Walk Test (6MWT) is a sub-maximal exercise test used to assess aerobic capacity and functional mobility by measuring the distance covered by the subject over a flat 25-meter corridor in 6 minutes. Greater distance covered indicates a better result. The score will be obtained in meters.
Time to complete the Five Times Sit to Stand Test (FTSST) | The test will be conducted at baseline, after 6 weeks, and upon completion of the 12-week program.
  This test is used to assess leg strength, dynamic balance and functional mobility. Subjects are timed in seconds as they rise from and return to a chair (standard height, 43-45 cm) five times. The performance in the test is recorded in seconds. Faster completion times indicate better performance. Testing occurs at the program's start, after 6 weeks, and upon completion of the 12-week program.
Time to climb one flight of stairs | The test will be conducted at baseline, after 6 weeks, and upon completion of the 12-week program.
  This test evaluates leg strength and functional mobility by timing subjects as they climb an 11-step flight of stairs as quickly as possible. Each step is 16 centimeters in height and 33 centimeters in depth. Testing will occur at the program's start, after 6 weeks, and upon the completion of the 12-week program.
Functional Reach Test (FRT) | The test will be conducted at baseline, after 6 weeks, and upon completion of the 12-week program.
  The FRT test will be used to assess dynamic balance by measuring how far a participant can reach while maintaining a fixed base of support. Participants will stand adjacent to a wall and extend the arm that is closer to the wall as far as possible. The distance reached by the participant along a measuring tape affixed to the wall is measured in centimeters. Three trials will be performed, and the average of the last two trials will be calculated.
Timed Up & Go Test (TUG) | The The test will be conducted at baseline, after 6 weeks, and upon completion of the 12-week program.
  The TUG test will be used to assess dynamic balance and functional mobility by timing the subjects as they rise from a chair, walk 3 meters, turn around, walk back to the chair, and sit down. The test score will be recorded in seconds, with a shorter TUG time indicating better results.
Forced Vital Capacity (FVC) | The test will be conducted at baseline, after 6 weeks, and upon completion of the 12-week program.
  This measure will be obtained through spirometry test as part of pulmonary function assessment. It represents the largest amount of air the subject can forcefully exhale after taking the deepest possible breath. Test results will be reported in liters.
Forced Expiratory Volume in one second (FEV1) | The test will be conducted at baseline, after 6 weeks, and upon completion of the 12-week program.
  This measure will be obtained through a spirometry test as part of pulmonary function assessment. It represents the maximum amount of air that the subject can force out his lungs in 1 second following maximal inhalation. Test results will be reported in liters.
Adherence to home-based program | From enrollment to the end of treatment at 12 weeks
  Adherence to the home-based exercise program will be calculated as a percentage out of the total number of exercises provided during a 12-week program (36 exercises in total).

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israek, Israel

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR